CLINICAL TRIAL: NCT00424385
Title: Phase I Study Investigating the Safety and Feasibility of Combining Imatinib Mesylate (Gleevec) With Sorafenib in Patients With Androgen-Independent Chemotherapy-Failure Prostate Cancer.
Brief Title: Study Combining Imatinib Mesylate (Gleevec) With Sorafenib in Patients With Androgen-independent Prostate Cancer (AIPC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncology Specialists, S.C. (Other)
Responsible Party: Principal Investigator, Dr. Sigrun Hallmeyer, Principal Investigator, Oncology Specialists, S.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CST1571BUS260 (0617)
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Prostate Cancer
Keywords: AIPC, Prostate cancer; prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Imatinib Mesylate; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Only 1 arm for the study - this arm gets both drugs, gleevec and sorafenib
  Interventions: Drug: Gleevec + Sorafenib

INTERVENTIONS:
Drug: Gleevec + Sorafenib — 400 mg Sorafenib every day (QD) 300mg Gleevec QD
  Other Names: Imatinib mesylate; Nexavar

SUMMARY:
Eligible patients will be enrolled in one of 4 cohorts where each cohort will allow 3 patients to be on study. Patients will receive both study drugs on escalated dosing schedule until the maximum of 400 mg PO BID is reached for both drugs or toxicity is established. Once the pre-specified 400 mg by mouth two times a day (PO BID) dosing for both drugs is reached without toxicity, the study will close for accrual. If toxicity is noted prior to reaching the 400 mg PO BID dosing, then the dosing schedule that is deemed safest as per study design will be the one used for any future phase II study.

DETAILED DESCRIPTION:
Gleevec and Sorafenib have modest efficacy in androgen-independent prostate cancer (AIPC) and the fact that both agents can be given orally with what appears to be tolerable side effects, we hypothesize that combining both agents may provide patients with another effective regimen in a disease where therapeutic options are limited. This study is designed to investigate the safety of combining Gleevec and Sorafenib as well as feasibility in AIPC patients who have failed one or more lines of systemic chemotherapy. Once safety is established, a follow-up phase II study will commence to investigate efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older.
2. Histologically documented diagnosis of Prostate Cancer regardless of Gleason score.
3. Androgen-Independent Prostate Cancer
4. At least one measurable site of disease
5. Patients must have failed one or more lines of systemic chemotherapy, regardless of the chemotherapeutic agent used. There is NO limit to how many lines of chemotherapy a patient can receive
6. Patients receiving anti-coagulation treatment with an agent such as heparin may be allowed to participate. Patients on Warfarin are NOT allowed to participate.
7. Last chemotherapy exposure 4 weeks prior to study entry
8. Prior exposure to Sorafenib is allowed as long as last Sorafenib dose was 3 weeks or more from study entry
9. Prior exposure to Gleevec is an EXCLUSION
10. Progression after chemotherapy can be demonstrated radiographically (as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria) or biochemically with prostate-specific antigen (PSA) being elevated more than 25% than previous value as long as a repeat PSA confirms progression. (repeat PSA should be done within 3 weeks from the last one). Patients with bone-only disease are considered progressing if there are two more lesions on a new bone scan.
11. Performance status 0,1, 2 (ECOG)
12. Adequate end organ function, defined as the following:

    * total bilirubin < 1.5 x Upper Limit of Normal (ULN), serum glutamate oxaloacetate transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) < 2.5 x Upper Limit of Normal (UNL), creatinine < 1.5 x Upper Limit of Normal (ULN), absolute neutrophil count (ANC) > 1.0 x 109/L, platelets > 75 x 109/L.
13. Men of childbearing potential must agree to employ an effective barrier method of birth control prior to the study entry, throughout the duration of the study and for up to 3 months following discontinuation of study drug.
14. Written, voluntary informed consent.
15. Patients are allowed the following concurrent therapies:

    * Intravenous bisphosphonates if administered for bone metastases
    * luteinizing hormone releasing hormone (LHRH) analogues
    * Narcotic-type medical interventions to control malignancy-related pain

Exclusion Criteria:

1. Patient has received any other investigational agents within 21 days of first day of study drug dosing, unless the disease is rapidly progressing.
2. Patient is < 3 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal or squamous cell skin cancer. Existence of any other malignant disease is not allowed.
3. Patient with Grade III/IV cardiac problems
4. Patient has a severe and/or uncontrolled medical disease
5. Patient has a known brain metastasis.
6. Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
7. Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
8. Pulmonary hemorrhage/bleeding event > Common Toxicity Criteria for Adverse Effects (CTCAE) Grade 2 within 4 weeks of first dose of study drug.
9. Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
10. Serious non-healing wound, ulcer, or bone fracture.
11. Use of St. John's Wort or rifampin (rifampicin).
12. Any condition that impairs patient's ability to swallow whole pills.
13. Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
14. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
15. Patient previously received radiotherapy to ³ 25 % of the bone marrow
16. Patient had a major surgery within 2 weeks prior to study entry.
17. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Nabhan, MD, Principal Investigator — Oncology Specialists, SC
Locations (2):
- United States (2):
  - Oncology Specialists, S.C, Niles, Illinois
  - Oncology Specialists, S.C, Park Ridge, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 patients were enrolled from our practice.
Pre-assignment Details: Patients enrolled failed previous chemotherapy.
Groups:
- Imatinib + Sorafenib: Both drugs, Gleevec + Sorafenib are given to all patients on study. There are 4 potential cohorts. Each will enroll 3 evaluable (patients that complete 2 cycles of treatment) patients. If a Dose Limiting Toxicity is demonstrated in a cohort, an additional 3 evaluable patients can be enrolled in that cohort.
  Cohort 0 was 400mg Sorafenib every day (QD)and 300mg of Imatinib QD. Cohort 1 was 400mg Sorafenib two times a day and 300mg QD Imatinib.
Period: Cohort 0
Arm/Group | Imatinib + Sorafenib
Started | 12
Completed | 6
Not Completed | 6
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 1
Period: Cohort 1
Arm/Group | Imatinib + Sorafenib
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Dose Limiting Toxicities (DLT's)
Description: Eligible patients were enrolled in one of 4 cohorts, where each cohort allowed 3 evaluable patients to be on study, patients withdrawn from treatment for reasons other than toxicity were not considered evaluable. If one of the three evaluable patients experienced a dose limiting toxicity (DLT) the cohort was expanded to 6 evaluable patients. Patients will receive both study drugs on escalated dosing schedule until the maximum of 400 mg PO BID is reached for both drugs or toxicity is established. If 2 out of six evaluable patients experience a dose limiting toxicity this would show that the Maximum Tolerated Dose (MTD) was the dose from the prior cohort.
Time Frame: up to 20 weeks
Population: Cohort 0: 6 evaluable patients were enrolled. Patients who withdrew for reasons other than toxicity were not considered evaluable for MTD. 1 out of 6 patients had a DLT, therefore Cohort 1 was started. Cohort 1: 2 DLTs were demonstrated from 5 evaluable patients. By definition the Maximum tolerated dose was the dosing schedule used in cohort 0.
Measure: Number; unit: participants
Groups:
- Imatinib + Sorafenib Cohort 0: 300mg every day (QD)Imatinib + 400mg every day (QD) Sorafenib, by mouth
- Imatinib + Sorafenib Cohort 1: 300mg every day (QD) Imatinib + 400mg twice daily (BID)Sorafenib, by mouth
Arm/Group | Imatinib + Sorafenib Cohort 0 | Imatinib + Sorafenib Cohort 1
Number analyzed (Participants) | 6 | 5
participants | 1 | 2

2. Secondary Outcome: Overall Clinical Benefit
Description: Overall Clinical Benefit was measured as the sum of complete response (CR), partial response (PR), and stable disease (SD).
Time Frame: up to 20 weeks
Population: There were 17 patients enrolled. 10 were evaluable for assessment of overall clinical benefit. 7 were not evaluable due to having received <1 cycle of drug.
Measure: Number; unit: percentage of evaluable participants
Groups:
- Imatinib + Sorafenib Cohort 0 & 1: Only 1 arm for the study - this arm gets both drugs, gleevec and sorafenib
Arm/Group | Imatinib + Sorafenib Cohort 0 & 1
Number analyzed (Participants) | 10
percentage of evaluable participants | 20

3. Secondary Outcome: Time to Disease Progression (TTP)
Description: Medium TTP is 2 months (range 1-5). 10 patients were evaluable for disease progression for these patients occurred between 1-5 months after starting the study. The TTP was calculated per protocol. For radiographic assessment Response Evaluation Criteria in Solid Tumors (RECIST) was used. Complete response = disappearance of all lesions. Partial response (PR)=30% or greater decrease in sum of longest diameter of measureable lesions SD. Lesions have no sufficient decrease for progressive disease and no sufficient increase to meet Progressive Disease (PD). PD more than 20% increase in sum of longest diameter of measurable lesions or 2 or more new bone mets. prostate-specific antigen (PSA) assessment for patients with measurable disease, PSA progression in the absence of measurable disease progression will not be considered progressive disease.
Time Frame: up to 5 cycles, an average of 20 weeks, from the day of first treatment until the date of the last dose of study drug
Measure: Median (Full Range); unit: months
Arm/Group | Imatinib + Sorafenib Cohort 0 & 1
Number analyzed (Participants) | 10
months | 2 [1 to 5]

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 6/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=17)
Broken C2 verebrae (Musculoskeletal and connective tissue disorders) | 1
Pain (General disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Urinary Tract Infection (Renal and urinary disorders) | 1
Chest pain (Cardiac disorders) | 1
Syncopal episode (Cardiac disorders) | 1
Dehydration (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Weakness (General disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Syndrome of Inappropriate Antiduretic Hormone (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=17)
Anemia (Blood and lymphatic system disorders) | 10
Appetite decreased (Gastrointestinal disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Albumin Low (Gastrointestinal disorders) | 8
Bruises easily (General disorders) | 1
Alopecia (General disorders) | 3
Anxiety (Psychiatric disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Alkaline Phosphatase (Hepatobiliary disorders) | 5
AST increased (Hepatobiliary disorders) | 4
Bilirubin increased (Renal and urinary disorders) | 2
Chest Pain (Cardiac disorders) | 1
Chloride Low (General disorders) | 3
Chills (General disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine Increased (Renal and urinary disorders) | 4
Alt Increased (Hepatobiliary disorders) | 1
Eyes tearing (Eye disorders) | 2
Edema lower extremity (General disorders) | 2
Edema periorbital (General disorders) | 1
Edema ankle (General disorders) | 1
Ear sore (Ear and labyrinth disorders) | 1
Fatigue (General disorders) | 7
Foot pain (Musculoskeletal and connective tissue disorders) | 1
Fever (Infections and infestations) | 2
Fall (General disorders) | 1
Desquamation (Skin and subcutaneous tissue disorders) | 6
Diarrhea (Gastrointestinal disorders) | 8
Dehydration (Gastrointestinal disorders) | 4
Dyspnea on Excertion (Respiratory, thoracic and mediastinal disorders) | 3
Depression (Psychiatric disorders) | 1
Hypotension (Cardiac disorders) | 1
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 3
Hypokalemia (Gastrointestinal disorders) | 2
Hypercalcemia (Gastrointestinal disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hypocalcemia (Gastrointestinal disorders) | 10
Hyperkalemia (Gastrointestinal disorders) | 4
Hyponatremia (Gastrointestinal disorders) | 4
Hot Flashes (General disorders) | 1
Hyperglycemia (Endocrine disorders) | 3
Insomnia (General disorders) | 2
Itching (Skin and subcutaneous tissue disorders) | 3
Infection (Infections and infestations) | 2
Leukopenia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 6
Libido decreased (Reproductive system and breast disorders) | 1
Muscle Pain (Musculoskeletal and connective tissue disorders) | 2
Mouth Dry (Gastrointestinal disorders) | 2
Mucositis (Gastrointestinal disorders) | 1
Magnesium decreased (Gastrointestinal disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Neuropathy (Musculoskeletal and connective tissue disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Oral candidiasis (Gastrointestinal disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 1
Pain (General disorders) | 6
Phosphorus High (Gastrointestinal disorders) | 1
Photo Sensitivity (Skin and subcutaneous tissue disorders) | 2
Total Protein Decreased (Gastrointestinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes